CLINICAL TRIAL: NCT01561508
Title: Double Blinded, Placebo Controlled Trial on the Effect of GABA Supplementation in the Progression of Type 1 Diabetes in Children
Brief Title: Effect of GABA Supplementation in the Progression of Type 1 Diabetes in Children
Acronym: GABA
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Unable to obtain IND currently
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Penny Jester, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UAB-GABA
Record Dates: First submitted 2012-03-16; First posted 2012-03-23 (Estimated); Last update posted 2012-12-24 (Estimated); Status verified 2012-12

CONDITIONS: Diabetes Mellitus
Keywords: diabetes mellitus; children
MeSH Terms: conditions — Diabetes Mellitus | interventions — gamma-Aminobutyric Acid; Xylitol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- GABA (Experimental): 2/3 of participants will be randomized to the GABA treatment group. Dosage will be based on body weight and will be adjusted at each study visit.
  Interventions: Drug: gamma-amino-butyric acid
- Placebo (Placebo Comparator): 1/3 of participants will receive placebo.
  Interventions: Dietary Supplement: Xylitol

INTERVENTIONS:
Drug: gamma-amino-butyric acid — gamma-amino butyric acid will be administered orally at a dose of 80mg/kg/day divided BID for one year.
  Other Names: GABA
  Arms: GABA
Dietary Supplement: Xylitol — The placebo group will be provided Xylitol powder dosed per body weight. Participants will be instructed to take powder orally twice a day for one year.
  Arms: Placebo

SUMMARY:
Type 1 diabetes mellitus (T1DM) is an autoimmune disease in which the body's immune system attacks and destroys the insulin producing beta cells of the pancreas. This condition is very prevalent, affecting up to 1:400/500 persons worldwide. Type 1 diabetes, previously known as juvenile diabetes, usually strikes in childhood, adolescence, or young adulthood, but lasts for a lifetime. To date, there have been no treatments that can arrest or reverse the ongoing beta cell destruction. The patients affected by this disease require multiple daily insulin injections to manage their blood sugars and usually have trouble regulating their blood sugars. Moreover, they are at risk for heart disease, kidney failure, eye problems, and other complications from this life-long condition.

The investigators plan to utilize gamma-amino butyric acid (GABA) in children with newly diagnosed T1DM. This neurotransmitter is made in the brain from the amino acid glutamate with the aid of vitamin B6. There have been some recent studies in diabetic mice utilizing GABA to reverse inflammation on the pancreas and improve hyperglycemia. GABA studied in healthy human subjects demonstrated that large oral doses of GABA increased insulin secretion from the pancreas.

The investigators propose that GABA given to children with new onset T1DM will be able to increase insulin production, suppress glucagon release, and decrease the inflammation surrounding the pancreas. The investigators hope this will at least prolong the beta cell life after diagnosis, if not lead to a cure for type 1 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Positive for any of the 3 measured antibodies GAD-65, ICA-512, or islet cell
* Must meet the ADA criteria for diabetes diagnosis
* Within 12 weeks of diagnosis of DMI at enrollment
* Peak stimulated c peptide of > 0.2 ng/mL with Mixed Meal Tolerance Test
* If post-menarchal they must use 2 forms of contraception during the study: this may include OCPs, abstinence and barrier methods. Abstinence will be accepted as a single method if used prior to enrollment.

Exclusion Criteria:

* Chronic systemic use of steroids
* Pregnancy or breastfeeding
* Seizure disorder
* Current use of Baclofen, Valium, Acamprosate, Neurontin, or Lyrica
* History of alcoholism/alcohol use
* Current use of anti diabetes drugs other than insulin
* Diagnosis of hemoglobinopathy
* Diagnosis of liver disease, cancer, cystic fibrosis, or renal failure

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2012-06; Primary Completion 2013-04 (Estimated)

PRIMARY OUTCOMES:
change in stimulated c-peptide | over 1 year
  We will measure c-peptide levels stimulated by a mixed meal tolerance test at baseline, six months and 12 months.

SECONDARY OUTCOMES:
change in HbA1C | over 1 year
  We will assess the change in hemoglobin A1C at baseline and every 3-4 months for a total duration of 1 year.
change in total daily insulin dose per kilogram | over 1 year
  We will assess the change in total daily insulin dose per kilogram of subject body weight at baseline and every 3-4 months for a total duration of 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Alison J Lunsford, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States